CLINICAL TRIAL: NCT00501137
Title: A Controlled Trial to Assess the Immunogenicity of a Proposed Paediatric Dosing Schedule of Human Papillomavirus Vaccine
Acronym: BCGov-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Simon Dobson (Other)
Collaborators: Ministry of Health, British Columbia (Other Government)
Responsible Party: Sponsor-Investigator, Simon Dobson, Associate Clinical Professor, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H07-00928
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Cervical Cancer; Genital Warts
Keywords: HPV; HPV vaccine; Gardasil; Human Papillomavirus; vaccine; 2 dose versus 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata | interventions — Papillomavirus Vaccines; Vaccines; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 16-26 year olds 3 doses HPV Vaccine (Active Comparator): Group 3 - 16-26 year olds receiving 3 doses HPV (Human Papillomavirus) Vaccine at 0, 2, 6 mths
  Interventions: Biological: HPV (Human Papillomavirus) Vaccine
- 3 dose 9-13 HPV Vaccine (Active Comparator): Group 2 - 9-13 year olds receiving 3 doses HPV (Human Papillomavirus) Vaccine at 0,2,6 mths
  Interventions: Biological: HPV (Human Papillomavirus) Vaccine
- 2 dose 9-13 yrs HPV Vaccine (Active Comparator): Group 1 9-13 year olds 2 doses HPV (Human Papillomavirus) Vaccine at 0 and 6 mths
  Interventions: Biological: HPV (Human Papillomavirus) Vaccine

INTERVENTIONS:
Biological: HPV (Human Papillomavirus) Vaccine — HPV (Human Papillomavirus) Vaccine received by all participants in groups 1, 2 and 3 according to the arm
  Other Names: Gardasil; Q-HPV; HPV Vaccine

SUMMARY:
Primary objective is to determine if antibody responses to HPV types 16 & 18 are non-inferior after a 2-dose paediatric regimen as compared to a 3-dose adult regimen of Q-HPV vaccination, with responses measured at Month 7.

DETAILED DESCRIPTION:
Human Papillomavirus (HPV) infection is a cause of cervical cancer. Immunogenicity, safety and efficacy in the prevention of persistent infection from HPV 16 and 18 has been proven using a 3-dose regimen in adolescent and adult females using the Quadrivalent Human Papillomavirus (Q-HPV) vaccine. The intensity of the immune response is inversely proportional to age. Immunogenicity in adolescents 9-15 years of age is 1.7 - 2 times greater than in 16-26 year old vaccine recipients. Paediatric dosing studies are necessary and prudent given limited provincial funding for new biologics acquisition and programme service delivery. A reduction from an adult 3-dose HPV vaccine regimen to a pediatric 2-dose regimen will result in increased compliance to the full vaccine series and in significant savings to the health care system both in the cost of biologics and of program delivery and administration.

ELIGIBILITY:
Inclusion Criteria:

* A female between, and including, 9-13 years (before 14th birthday) and 16-26 years of age (before 27th birthday) at the time of the first vaccination.
* Healthy
* Not pregnant
* Four or less sexual partners over lifetime as reported by subject. (Sexual activity is defined as intercourse)
* Not planning to become pregnant or likely to become pregnant
* No reported history of genital warts
* No laboratory confirmed history of cervical intraepithelial neoplasia
* No previous vaccination against HPV
* No administration of immunoglobulin and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period
* No previous anaphylactic reaction to HPV vaccine or any vaccine related component including aluminum hydroxyphosphate sulfate and polysorbate 80
* No confirmed or suspected immunosuppressive or immunodeficient condition based on medical history
* No bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
* Cannot be already enrolled in any clinical trial in which investigational vaccine or drug are being administered

Exclusion Criteria

* Pregnant
* Female planning to become pregnant or likely to become pregnant (as determined by the investigator) during the study duration Part 1 (0-7 months)
* Reported history of genital warts
* Laboratory confirmed history of cervical intraepithelial neoplasia
* Greater than four lifetime sexual partners involving sexual intercourse
* Previous vaccination against HPV
* Administration of immunoglobulin and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period
* A previous anaphylactic reaction to HPV vaccine or any vaccine related component including aluminum hydroxyphosphate sulfate and polysorbate 80
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history (e.g. HIV infection, genetic defect, immunosuppressive therapy). *Chronic administration (defined as more than 14 days) of immune-modifying drugs within 6 months prior to the first vaccine dose or planned use during the study period is exclusionary (corticosteroid use - immune-modifying level is ≥0.5 mg/kg/day; inhaled or topical steroids are acceptable).
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection (thrombocytopaenia, coagulation disorder, anti-coagulant therapy).
* Enrollment in any clinical trial in which investigational vaccine or drug are being administered

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 830 (Actual)
Dates: Start 2007-07; Primary Completion 2008-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Primary Objective Part 1 | Measured after Month 7
  To determine if antibody responses to HPV types 16 & 18 are non-inferior after a 2-dose paediatric regimen as compared to a 3-dose adult regimen of Q-HPV vaccination
Primary Objective Part 2 | At 18, 24 and 36mths post dose 1
  To compare the serum antibody responses to HPV 6, 11, 16 & 18 at months 18, 24 and 36 in 2-dose adolescent arm, 3-dose adolescent arm and 3-dose adult arm of the study.
Primary Objective Part 2 | Measured at 36 mths
  To evaluate the memory B cell and T helper cell mediated immune response to Q-HPV vaccine in the 2-dose adolescent, 3-dose adolescent and 3-dose adult arms

SECONDARY OUTCOMES:
Secondary Objective Part 1 & 2 - Antibody responses 2 doses between 9-13 vs 16-26 | Measured at 7, 18,24 and 36 mths
  To demonstrate that 2-doses of Q-HPV vaccine administered to 9-13 year old females produces a serum antibody response to HPV 6 and 11 that is similar to the response seen in 16-26 year olds
Secondary Objective Part 1 & 2 - HPV 16 and 18 2 doses versus 3 | Measured at 7,18,24 and 36 mths
  To evaluate the antibody responses to HPV 16 and 18 in 9-13 year old females after a 2-dose versus a 3-dose Q-HPV regimen
Secondary Objective Part 1 seroconversion rates | Measured at 7 mths
  To evaluate seroconversion rates to HPV 6, 11, 16, and 18
Secondary Objective Part 1 Memory Response | Measured at 7 mths
  To evaluate the memory B cell and T helper cell mediated immune response to Q-HPV vaccine in the 2-dose adolescent, 3-dose adolescent and 3-dose adult arms

CONTACTS AND LOCATIONS:
Overall Officials: Simon Dobson, MD, Principal Investigator — University of British Columbia; David Scheifele, MD, Study Director — Vaccine Evaluation Centre, Vancouver; Meena Dawar, MD, Study Director — Vaccine Evaluation Centre, Vancouver; Tobias Kollman, MD, Study Director — Vaccine Evaluation Centre, Vancouver; Shelly McNeil, MD, Study Director — Centre for Vaccinology, Halifax; Scott Halperin, MD, Study Director — Centre for Vaccinology, Halifax; Joanne Langley, MD, Study Director — Centre for Vaccinology, Halifax; Marc Dionne, MD, Study Director — Centre de Recherche du CHUL (CHUQ), Quebec
Locations (1):
- Vaccine Evaluation Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Dobson SR, McNeil S, Dionne M, Dawar M, Ogilvie G, Krajden M, Sauvageau C, Scheifele DW, Kollmann TR, Halperin SA, Langley JM, Bettinger JA, Singer J, Money D, Miller D, Naus M, Marra F, Young E. Immunogenicity of 2 doses of HPV vaccine in younger adolescents vs 3 doses in young women: a randomized clinical trial. JAMA. 2013 May 1;309(17):1793-802. doi: 10.1001/jama.2013.1625. PMID 23632723
- [Result] Krajden M, Cook D, Yu A, Chow R, Su Q, Mei W, McNeil S, Money D, Dionne M, Palefsky J, Karunakaran K, Kollmann T, Ogilvie G, Petric M, Dobson S. Assessment of HPV 16 and HPV 18 antibody responses by pseudovirus neutralization, Merck cLIA and Merck total IgG LIA immunoassays in a reduced dosage quadrivalent HPV vaccine trial. Vaccine. 2014 Jan 23;32(5):624-30. doi: 10.1016/j.vaccine.2013.09.007. Epub 2013 Sep 19. PMID 24055350
- [Result] Krajden M, Cook D, Yu A, Chow R, Mei W, McNeil S, Money D, Dionne M, Karunakaran KP, Palefsky JM, Dobson S, Ogilvie G, Petric M. Human papillomavirus 16 (HPV 16) and HPV 18 antibody responses measured by pseudovirus neutralization and competitive Luminex assays in a two- versus three-dose HPV vaccine trial. Clin Vaccine Immunol. 2011 Mar;18(3):418-23. doi: 10.1128/CVI.00489-10. Epub 2011 Jan 19. PMID 21248158
- [Result] Smolen KK, Gelinas L, Franzen L, Dobson S, Dawar M, Ogilvie G, Krajden M, Fortuno ES 3rd, Kollmann TR. Age of recipient and number of doses differentially impact human B and T cell immune memory responses to HPV vaccination. Vaccine. 2012 May 21;30(24):3572-9. doi: 10.1016/j.vaccine.2012.03.051. Epub 2012 Mar 31. PMID 22469863
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: click here for study details — http://www.vec.med.ubc.ca